CLINICAL TRIAL: NCT01653379
Title: A Phase 2A, Open-label, Dose-ranging and Pharmacokinetic Study of an Oral Vitamin D Compound (DP001) in Secondary Hyperparathyroidism in Patients on Hemodialysis
Brief Title: A Phase 2A Dose-ranging and Pharmacokinetic Study of an Oral Vitamin D Compound (DP001) in Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deltanoid Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2MD-7H-2A
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DP001 (Experimental): DP001 softgel capsules; 55 ng to 550 ng per dose, administered 3 times weekly for 4 weeks
  Interventions: Drug: DP001

INTERVENTIONS:
Drug: DP001 — DP001 softgel capsules; 55 ng to 550 ng per dose, administered 3 times weekly for 4 weeks

SUMMARY:
This is an open-label, dose-ranging study of the vitamin D analog DP001 in patients with end-stage renal disease (ESRD). The primary goals of this 4-week Phase 2A study are to identify an appropriate starting dose of DP001 to be used in subsequent studies in this population and for evaluation of pharmacokinetics of DP001 in ESRD patients.

DETAILED DESCRIPTION:
Vitamin D hormone or analogs, when bound to the vitamin D receptor, suppress PTH synthesis by binding to a negative regulatory element in the promoter of the PTH gene, and have been used successfully in the clinic to reduce elevated PTH levels in dialysis patients and other CKD patients. DP001 is a highly potent vitamin D compound.

In two clinical trials testing DP001 in postmenopausal women, oral DP001 reduced PTH levels in a dose-dependent manner, with a dose of 220 ng lowering PTH by at least 30% in a majority of patients following one or six months of daily dosing.

This study is an open-label, dose-ranging study of DP001 in ESRD patients with secondary hyperparathyroidism. Cohorts of up to 6 patients will be enrolled and administered oral DP001 at 110 ng three times per week for four weeks. Laboratory data from each cohort will be assessed and used to determine a dose for the next cohort. Up to 5 dose-ranging cohorts will be studied, with the goal of identifying an appropriate dose for a randomized, placebo-controlled study of oral DP001 for 12 weeks. The data will also be used to select an appropriate dose for an additional cohort of 12 open-label patients in the current study in which the pharmacokinetics of DP001 following a single dose and after repeated doses will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with ESRD and must be on hemodialysis 3 times per week for at least 3 months
* Plasma intact PTH value >/= 300 pg/mL

Exclusion Criteria:

* Currently taking drugs affecting vitamin D metabolism
* History of symptomatic ventricular dysrhythmias, congestive heart failure, angina pectoris, myocardial infarction, coronary angioplasty, or coronary artery bypass grafting
* Active malignancy
* Clinically significant liver disease
* Active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in intact parathyroid hormone levels in blood | Baseline and 4 weeks

SECONDARY OUTCOMES:
Blood levels of DP001 | Multiple time points following single dose and 4 weeks of dosing
  1, 2, 4, 8, 24, and 48 hours following a single dose; 1, 2, 4, 8, 24, 48, 72, and 96 hours following multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Thadhani, MD, Study Chair — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Tucson, Arizona
  - Tustin, California
  - Denver, Colorado
  - St Louis, Missouri
  - Greenville, Texas
  - Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here: — http://deltanoid.com/contact.php